CLINICAL TRIAL: NCT00808834
Title: Non-dispense Comfort Comparison of Two Silicone Hydrogel Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P-335-C-008
Record Dates: First submitted 2008-12-11; First posted 2008-12-16 (Estimated); Results first posted 2010-10-04 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Senofilcon A / Lotrafilcon A (Other): Senofilcon A, followed by Lotrafilcon A
  Interventions: Device: Lotrafilcon A contact lens; Device: Senofilcon A contact lens
- Lotrafilcon A / Senofilcon A (Other): Lotrafilcon A, followed by Senofilcon A
  Interventions: Device: Lotrafilcon A contact lens; Device: Senofilcon A contact lens

INTERVENTIONS:
Device: Lotrafilcon A contact lens — Investigational, silicone hydrogel, spherical, soft contact lens
Device: Senofilcon A contact lens — Commercially marketed, silicone hydrogel, spherical, soft contact lens

SUMMARY:
The purpose of this study is to compare subjective responses to two contact lenses after 15 minutes of wear.

ELIGIBILITY:
Inclusion Criteria:

* Currently wearing soft contact lenses
* Replaces lenses on a weekly or longer schedule
* Other protocol-defined inclusion/exclusion criteria may apply

Exclusion Criteria:

* Requires concurrent ocular medication
* Eye injury or surgery within twelve weeks immediately prior to enrollment
* Currently wearing soft toric lens wearers
* Those who dispose of their soft lenses on a daily basis
* Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Senofilcon A / Lotrafilcon A | Lotrafilcon A / Senofilcon A
Started | 97 | 99
Completed | 97 | 99
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Senofilcon A / Lotrafilcon A | Lotrafilcon A / Senofilcon A
Started | 97 | 99
Completed | 97 | 99
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled and exposed subjects.
Arm/Group | Overall
Number analyzed (Participants) | 196
Age Continuous [Mean (Standard Deviation); unit: years] | 30.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 55
Region of Enrollment [Number; unit: participants]
  United States | 196

OUTCOME MEASURES:

1. Primary Outcome: Comfort After Insertion
Description: Evaluated by the subject and measured on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 30-60 seconds after initial insertion
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Scale 1-10
Groups:
- Senofilcon A: Commercially marketed, silicone hydrogel, spherical, soft contact lens
- Lotrafilcon A: Investigational, silicone hydrogel, spherical, soft contact lens
Arm/Group | Senofilcon A | Lotrafilcon A
Number analyzed (Participants) | 193 | 193
Scale 1-10 | 8.7 (1.5) | 7.7 (2.4)

ADVERSE EVENTS:
Time Frame: 30 days, duration of the trial.
Description: Subjects wore 2 pairs of contact lenses, 15 minutes per pair.
Arm/Group | Senofilcon A | Lotrafilcon A
Serious Adverse Events (participants affected / at risk) | 0/196 | 0/196
Other Adverse Events (participants affected / at risk) | 0/196 | 0/196

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.